CLINICAL TRIAL: NCT02215291
Title: High Resolution Optical Imaging of the Esophagus Using the NvisionVLE™ Imaging Registry
Brief Title: NvisionVLE™ Registry System Registry
Status: Completed | Type: Observational
Sponsor: NinePoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 13_02
Record Dates: First submitted 2014-07-31; First posted 2014-08-13 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Esophagogastroduodenoscopy
Keywords: Undergoing Esophagogastroduodenoscopy (EGD) or endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing EGD or esophagoscopy: The cohort includes patients undergoing EGD or esophagoscopy for initial diagnosis or initial staging and mapping, surveillance of non-treated disease, and treatment (initial or ongoing) or post-treatment surveillance

SUMMARY:
Prospective, multi-site registry with longitudinal follow up for patients undergoing EGD or endoscopy. The primary objective is to provide a collection of patient NvisionVLE™ procedural data for participating physicians, including, but not limited to, imaging data, clinical utility data, demographics, pathology, treatment, and surveillance.

DETAILED DESCRIPTION:
This is a prospective, multi-site registry with longitudinal follow up for patients undergoing EGD or endoscopy. The primary objective is to provide a collection of patient NvisionVLE™ procedural data for participating physicians, including, but not limited to, imaging data, clinical utility data, demographics, pathology, treatment, and surveillance.

Up to 1000 patients from up to 20 sites nationwide.

There are no protocol defined follow up visits. Patients will undergo an initial baseline Volumetric Laser Endomicroscopy (VLE) procedure. A patient with a negative screening examination may not require additional screening endoscopies. For patients with established disease, further surveillance endoscopies will vary based on the extent of the disease (e.g. every 3 months, every 6 months, annual), which is based on the following American Society for Gastrointestinal Endoscopy (ASGE) guideline: the role of endoscopy in the surveillance of premalignant conditions of the upper GI tract. If patients have additional VLE procedures during the enrollment period, associated data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for an endoscopic examination of the esophagus
* Ability to provide written, informed consent to participate in the Registry

Exclusion Criteria:

* Patients for whom use of the NvisionVLE device would be in conflict with the Instructions for Use (IFU)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 20 sites; each site will have the opportunity to enroll up to 100 patients. There will be up to 1000 patients enrolled in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Percent of patients with endoscopically visible disease/ suspicious areas as determined by the physician | Baseline
  No protocol defined follow up visits. Patients will undergo an initial baseline Volumetric Laser Endomicroscopy (VLE) procedure. If patients have additional VLE procedures during the enrollment period, associated data will be collected.
Percent of patients with VLE visible abnormalities/ suspicious areas as determined by the physician | Baseline
  No protocol defined follow up visits. Patients will undergo an initial baseline VLE procedure. If patients have additional VLE procedures during the enrollment period, associated data will be collected.
Percent of patients with histologically confirmed disease and a breakdown of diseases observed | Baseline
  No protocol defined follow up visits. Patients will undergo an initial baseline VLE procedure. If patients have additional VLE procedures during the enrollment period, associated data will be collected.
Percent of treated patients with endoscopic and VLE identified areas of retained or persistent abnormalities at the first endoscopic evaluation after treatment | Baseline
  No protocol defined follow up visits. Patients will undergo an initial baseline VLE procedure. If patients have additional VLE procedures during the enrollment period, associated data will be collected.
Percent of treated patients undergoing surveillance with endoscopic and VLE areas of recurrent abnormality diagnosed by histology as disease | Baseline
  No protocol defined follow up visits. Patients will undergo an initial baseline VLE procedure. If patients have additional VLE procedures during the enrollment period, associated data will be collected.
Percent of patients with abnormalities/ suspicious areas identified by the physician as subsquamous visualized on VLE and not seen on endoscopy | Baseline
  No protocol defined follow up visits. Patients will undergo an initial baseline VLE procedure. If patients have additional VLE procedures during the enrollment period, associated data will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Smith, MD, MBA, Principal Investigator — Temple University Hospital
Locations (18):
- United States (18):
  - Univeristy of South Alabama, Mobile, Alabama
  - University of Southern California, Los Angeles, California
  - University of California Irvine, Orange, California
  - Mayo Clinic, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Ochsner Health System, Kenner, Louisiana
  - VA Boston Health Care System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - North Shore/ LIJ, Long Island City, New York
  - Weill Cornell Medical College/NewYork-Presbyterian Hospital, New York, New York
  - Columbia Univeristy, New York, New York
  - Geisinger, Danville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- [Derived] Smith MS, Cash B, Konda V, Trindade AJ, Gordon S, DeMeester S, Joshi V, Diehl D, Ganguly E, Mashimo H, Singh S, Jobe B, McKinley M, Wallace M, Komatsu Y, Thakkar S, Schnoll-Sussman F, Sharaiha R, Kahaleh M, Tarnasky P, Wolfsen H, Hawes R, Lipham J, Khara H, Pleskow D, Navaneethan U, Kedia P, Hasan M, Sethi A, Samarasena J, Siddiqui UD, Gress F, Rodriguez R, Lee C, Gonda T, Waxman I, Hyder S, Poneros J, Sharzehi K, Di Palma JA, Sejpal DV, Oh D, Hagen J, Rothstein R, Sawhney M, Berzin T, Malik Z, Chang K. Volumetric laser endomicroscopy and its application to Barrett's esophagus: results from a 1,000 patient registry. Dis Esophagus. 2019 Nov 13;32(9):doz029. doi: 10.1093/dote/doz029. PMID 31037293